CLINICAL TRIAL: NCT01237847
Title: A Brief Intervention to Improve Adherence in Teens With Inflammatory Bowel Disease
Acronym: PHONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Medical College of Wisconsin (Other); Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Rachel Neff Greenley PhD, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CCFA#2838
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; IBD; Crohn's disease; ulcerative colitis; adolescent
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait List (Other)
  Interventions: Behavioral: Wait list comparison group
- 2 phone sessions (Experimental)
  Interventions: Behavioral: 2 Family-based problem solving phone sessions
- 4 phone sessions (Experimental)
  Interventions: Behavioral: 4 Family-based problem solving phone intervention sessions

INTERVENTIONS:
Behavioral: 2 Family-based problem solving phone sessions — 2 family-based problem solving phone sessions to address and ameliorate barriers to adherence.
  Arms: 2 phone sessions
Behavioral: 4 Family-based problem solving phone intervention sessions — 4 family-based problem solving phone sessions to address and ameliorate barriers to adherence.
  Arms: 4 phone sessions
Behavioral: Wait list comparison group — Wait list comparison group to receive intervention at later point.
  Arms: Wait List

SUMMARY:
This project will test if a phone intervention can improve the medicine-taking behavior of teens with IBD. The investigators will study teens who are taking medicine by mouth. The investigators will test if two phone calls that help teens solve problems with their IBD medicine help to increase how often teens take their medicine. The study will also see if there is any extra benefit of more sessions (four compared to two). The investigators will ask 90 teens to be in the study. Teens can be in the study if they are 11-18 years old and speak English. They must also take an IBD medication by mouth and have a parent who also wants to be in the study. Teens who agree to be in the study will fill out forms at the beginning (participant week 0), middle (participant week 12), and end of the study (participant week 20). After assessment 1, they will be randomly assigned to either receive 2 phone calls or a wait list group (participant weeks 6-10). After that, they will complete a second assessment. After the second assessment, teens who got the 2 phone calls right will be re-randomized to two more sessions or no more sessions (participant weeks 14-18). Teens who were in the wait list group will get two phone sessions (participant weeks 14-18). After that, there will be a final assessment (participant week 20). The investigators expect the phone intervention sessions to reduce barriers to medicine taking, improve medicine taking, and improve teen quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patient age 11-18 years
* patient English speaking
* patient legal guardian willing to participate
* patient on oral IBD maintenance medication for 3 months or longer

Exclusion Criteria:

* history of significant parent-reported cognitive or developmental delay

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Adherence | beginning at baseline - week 20
  participants will use MEMS bottles to capture adherence data from participant week 0 - participant week 20. Additionally, adherence interviews and pill counts will be conducted at participant week 0, 12, and 20.

SECONDARY OUTCOMES:
Quality of Life | at baseline, week 12, and week 20
Adherence barriers | at baseline, week 12, and week 20

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Neff Greenley, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Greenley RN, Gumidyala AP, Nguyen E, Plevinsky JM, Poulopoulos N, Thomason MM, Walter JG, Wojtowicz AA, Blank E, Gokhale R, Kirschner BS, Miranda A, Noe JD, Stephens MC, Werlin S, Kahn SA. Can You Teach a Teen New Tricks? Problem Solving Skills Training Improves Oral Medication Adherence in Pediatric Patients with Inflammatory Bowel Disease Participating in a Randomized Trial. Inflamm Bowel Dis. 2015 Nov;21(11):2649-57. doi: 10.1097/MIB.0000000000000530. PMID 26218142